CLINICAL TRIAL: NCT00005591
Title: Phase II Study of Anti-Epidermal Growth Factor Receptor (EGFr) Antibody C225 in Combination With Gemcitabine in Patients With Advanced Pancreatic Cancer
Brief Title: Cetuximab Plus Gemcitabine in Treating Patients With Locally Advanced, Metastatic, or Recurrent Cancer of the Pancreas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067696; UAB-9929; IMCL-CP02-9814; UAB-F990927003; NCI-G00-1729
Record Dates: First submitted 2000-05-02; First posted 2004-08-09 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cell from dividing so they stop growing or die. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cetuximab plus gemcitabine in treating patients who have locally advanced, metastatic, or recurrent cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine objective response, time to progression, survival, clinical benefit response, and quality of life of patients with locally advanced, metastatic, or recurrent adenocarcinoma of the pancreas when treated with cetuximab and gemcitabine. II. Determine the safety and toxicity profile of this regimen in this patient population.

OUTLINE: This is a multicenter study. Patients receive a test dose of cetuximab IV over 10 minutes followed by a 30 minute observation period. Following observation, patients receive a loading dose of cetuximab IV over 1-2 hours followed 1 hour later by gemcitabine IV over 30 minutes weekly for 7 weeks. Following 1 week of rest, patients with stable or responding disease continue treatment for a maximum of 6 months. During subsequent courses, patients receive maintenance doses of cetuximab IV over 1 hour weekly for 8 weeks. Gemcitabine IV is administered over 30 minutes weekly for 3 weeks, followed by 1 week of rest, and then repeated for a total treatment course of 8 weeks. Treatment continues in the absence of unacceptable toxicity or disease progression. Quality of life is assessed at baseline, after each course of therapy, and at 3 months after therapy. Patients are followed every 3 months until evidence of disease progression.

PROJECTED ACCRUAL: A minimum of 40 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed locally advanced, metastatic, or recurrent adenocarcinoma of the pancreas that is not amenable to curative surgical resection Immunohistochemical evidence of EGFr expression of 1+ or greater Measurable disease No history of treated or active brain metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Hemoglobin at least 9 g/dL Platelet count at least 100,000/mm3 No unstable coagulation disorders Hepatic: AST/ALT no greater than 5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 5 times ULN Bilirubin no greater than 2 times ULN Renal: Creatinine no greater than 2.5 mg/dL Cardiovascular: No uncontrolled hypertension or arrhythmias No unstable congestive heart failure Neurologic: No uncontrolled seizure disorder No active neurological disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No concurrent unstable medical condition (e.g., uncontrolled diabetes mellitus or active infections requiring systemic antibiotics, antivirals, or antifungals)

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior murine monoclonal antibody therapy No prior cetuximab Chemotherapy: No prior chemotherapy for advanced pancreatic cancer Prior adjuvant chemotherapy following complete surgical resection allowed provided cancer recurrence was first documented more than 6 months after completion of treatment Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior radiotherapy to only site of measurable disease unless documented disease progression since prior irradiation Surgery: Prior surgical resection allowed Other: At least 4 weeks since other prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-10; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert F. LoBuglio, MD, Study Chair — University of Alabama at Birmingham